CLINICAL TRIAL: NCT07141979
Title: Effects of tDCS on Cognitive Flexibility and EEG Oscillations in Orthorexia Nervosa
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Bahar Güntekin, Prof. Dr., Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: E-10840098-202.3.02-35.59
Record Dates: First submitted 2025-08-18; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-07

CONDITIONS: Orthorexia Nervosa
Keywords: Orthorexia Nervosa; cognitive flexibility; tDCS; EEG Oscillations
MeSH Terms: conditions — Orthorexia Nervosa

STUDY DESIGN:
Intervention Model Description: It is an experimental, randomised controlled trial. The data will be collected with the convenience sampling method from volunteer healthy people and individuals with orthorexia nervosa. The matched-group design method will be used.
Who Masked: Participant
Masking Description: Participants will not know that which group they will be in
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): Participants will take active tDCS stimulation
  Interventions: Device: Active tDCS
- Control group (Sham Comparator): Participants will take sham tDCS stimulation
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — 20 min, 2 milliampere (mA), Anodal tDCS in left DLPFC
  Arms: Experimental group
Device: Sham tDCS — 20 min, left DLPFC Sham tDCS
  Arms: Control group

SUMMARY:
Orthorexia Nervosa (ON); is a condition characterized by individuals being overly focused on healthy eating habits, constantly checking and classifying the foods they will consume. ON has not yet been clinically defined as an eating disorder or in a different category, and has not been included in DSM-5. Cognitive flexibility can be defined as a person's ability to quickly change their thinking and behaviors to adapt to different situations and changing conditions. It has been reported that cognitive flexibility skills are impaired in ON. There is evidence that tDCS, a neuromodulation method, increases cognitive flexibility skills. On the other hand, although there are EEG studies on eating disorders, there is no EEG study directly studying ON, and there is no information on the EEG profiles of individuals with high ON scores. For this reason, EEG studies on eating disorders and obsessive behaviors are generally generalized to orthorexia nervosa and are interpreted. This study aims to compare the EEG oscillations and cognitive flexibility skills of individuals with high ON scores with a control group and to examine the effects of anodal tDCS application on these two variables. For this purpose, a total of 48 individuals, 24 healthy and 24 high ON scores, will be included in the study. Participants will be randomly assigned to tDCS experimental and control groups. Therefore, 48 participants will be divided into 4 different subgroups of 12 people each. Data collection tools will be Informed Consent Form, Demographic Information Form, Beck Depression Inventory, Orthorexia Nervosa Test (TON-17), Cognitive flexibility task. First, participants will be subjected to a cognitive flexibility task by taking simultaneous EEG recordings, then tDCS stimulation will be initiated (active or sham) and after stimulation, a cognitive flexibility task will be performed by taking simultaneous EEG recordings again. EEG analyses will be performed using the Brain-Vision Analyzer program. Repeated Measures Analysis of Variance (within-group and between-groups) will be used in statistical analyses.

DETAILED DESCRIPTION:
Measurement instruments:

Informed Voluntary Consent Form Demographic Information Form Edinburgh Hand Preference Survey Beck Depression Scale Test of Orthorexia Nervosa (TON-17) Cognitive Flexibility Task EEG and tDCS devices Statistics: Statistical analyses will be conducted using SPSS 25.0 (Statistical Package for Social Sciences) for Windows, and EEG data will be analyzed using the Brain-Vision Analyzer software.

Descriptive statistics for group variables such as age and education will be presented as means and standard deviations, while gender will be reported as frequency and percentage.

The normality of the distribution of variables will be assessed using the Kolmogorov-Smirnov test, and appropriate parametric or non-parametric tests will be applied based on the results.

To evaluate pre-test and post-test data for cognitive flexibility and EEG measures in the experimental and control groups, Repeated Measures Analysis of Variance (within- and between-subjects) or its non-parametric equivalent, the Friedman Test, will be used.

For all statistical tests, a significance level of p < 0.05 will be considered as the threshold for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-40,
* Having a score of 17 or less on the Beck Depression Inventory
* Having a score of 61 or more on the Test for Orthorexia Nervosa (TON-17) for the orthorexia group

Exclusion Criteria:

* Having a history of serious neurological and psychiatric illness,
* Currently taking medication that alters the cortical excitability level,
* Having visual defects that cannot be corrected with glasses
* Use of intracranial metal objects, implanted stimulating devices or pacemakers

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in EEG Oscillations in individuals with Orthorexia Nervosa for active vs. sham stimulation | Baseline, 5 minutes after completion of the active/sham stimulation
  The EEG oscillations recording the event brain oscillations during the cognitive flexibility task from pre and post measurements. There are the five frequencies band which are Delta (0.5-3,5 Hz), Theta (4-7 Hz), Alpha (8-13 Hz), Beta (15-30 Hz) and Gamma (30-100 Hz). Data will be record simultaneously and analyzed. The analysis will be done with the BrainVisionAnalyzer program and power analysis will be made in Delta, Theta, Alpha, Beta, Gamma bands and the averages will be compared. Oscillations will be evaluated in terms of averages changing as an indicator of the effect of the neuromodulation preceding it.
Change in Cognitive Flexibility Task score in individuals with Orthorexia Nervosa for active vs. sham stimulation | Baseline, 20 minutes after completion of the active/sham stimulation
  A structured task-switching paradigm will be used to measure cognitive flexibility skills from pre and post test score in individuals with Orthorexia Nervosa
  * The paradigm consists of two conditions: trials with a task switch and trials without a task switch. The experiment will include two blocks, with a total of 320 trials. Each block will contain 160 phases, consisting of 80 trials with a task switch and 80 trials without a task switch. Score averages will compare between pre and post test. Data will be record Excel by Psychopy program simultaneously. Performance will be evaluated for accuracy as an indicator of the effect of the neuromodulation preceding it.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Emek Savas DD, Yerlikaya D, G Yener G, Oktem Tanor O. Validity, Reliability and Normative Data of the Stroop Test Capa Version. Turk Psikiyatri Derg. 2020 Spring;31(1):9-21. doi: 10.5080/u23549. English, Turkish. PMID 32594475
- [Background] Du M, Peng Y, Li Y, Zhu Y, Yang S, Li J, Zou F, Wang Y, Wu X, Zhang Y, Zhang M. Effect of trait anxiety on cognitive flexibility: Evidence from event-related potentials and resting-state EEG. Biol Psychol. 2022 Apr;170:108319. doi: 10.1016/j.biopsycho.2022.108319. Epub 2022 Mar 22. PMID 35331781
- [Background] Dong G, Wang Y, Chen X. Anodal occipital tDCS enhances spontaneous alpha activity. Neurosci Lett. 2020 Mar 16;721:134796. doi: 10.1016/j.neulet.2020.134796. Epub 2020 Jan 30. PMID 32006627
- [Background] Donaldson PH, Kirkovski M, Yang JS, Bekkali S, Enticott PG. High-definition tDCS to the right temporoparietal junction modulates slow-wave resting state power and coherence in healthy adults. J Neurophysiol. 2019 Oct 1;122(4):1735-1744. doi: 10.1152/jn.00338.2019. Epub 2019 Aug 28. PMID 31461371
- [Background] Darna M, Stolz C, Jauch HS, Strumpf H, Hopf JM, Seidenbecher CI, Schott BH, Richter A. Frontal theta oscillations and cognitive flexibility: Age-related modulations in EEG activity. Aging Brain. 2025 Jun 24;8:100142. doi: 10.1016/j.nbas.2025.100142. eCollection 2025. PMID 40620518
- [Background] Chrysikou EG, Hamilton RH, Coslett HB, Datta A, Bikson M, Thompson-Schill SL. Noninvasive transcranial direct current stimulation over the left prefrontal cortex facilitates cognitive flexibility in tool use. Cogn Neurosci. 2013;4(2):81-9. doi: 10.1080/17588928.2013.768221. PMID 23894253
- [Background] Cavinato M, Genna C, Formaggio E, Gregorio C, Storti SF, Manganotti P, Casanova E, Piperno R, Piccione F. Behavioural and electrophysiological effects of tDCS to prefrontal cortex in patients with disorders of consciousness. Clin Neurophysiol. 2019 Feb;130(2):231-238. doi: 10.1016/j.clinph.2018.10.018. Epub 2018 Nov 29. PMID 30580246
- [Background] Borwick C, Lal R, Lim LW, Stagg CJ, Aquili L. Dopamine depletion effects on cognitive flexibility as modulated by tDCS of the dlPFC. Brain Stimul. 2020 Jan-Feb;13(1):105-108. doi: 10.1016/j.brs.2019.08.016. Epub 2019 Aug 31. PMID 31494070
- [Background] Berchio C, Annen LC, Bouamoud Y, Micali N. Temporal dynamics of cognitive flexibility in adolescents with anorexia nervosa: A high-density EEG study. Eur J Neurosci. 2023 Mar;57(6):962-980. doi: 10.1111/ejn.15921. Epub 2023 Feb 7. PMID 36683346
- [Background] Alizadehgoradel J, Nejati V, Sadeghi Movahed F, Imani S, Taherifard M, Mosayebi-Samani M, Vicario CM, Nitsche MA, Salehinejad MA. Repeated stimulation of the dorsolateral-prefrontal cortex improves executive dysfunctions and craving in drug addiction: A randomized, double-blind, parallel-group study. Brain Stimul. 2020 May-Jun;13(3):582-593. doi: 10.1016/j.brs.2019.12.028. Epub 2020 Jan 3. PMID 32289681
- [Background] Aboulafia-Brakha T, Manuel AL, Ptak R. Prefrontal transcranial direct current stimulation facilitates affective flexibility. Neuropsychologia. 2016 Jun;86:13-8. doi: 10.1016/j.neuropsychologia.2016.03.030. Epub 2016 Mar 30. PMID 27039163